CLINICAL TRIAL: NCT04234035
Title: Shared Decision-Making for the Promotion of Patient-Centered Imaging in the Emergency Department: Suspected Kidney Stones
Brief Title: Shared Decision-Making for the Promotion of Patient-Centered Imaging in the ED: Suspected Kidney Stones
Acronym: ED-KSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Schoenfeld, MD, Assistant Professor, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BH-19-168
Record Dates: First submitted 2019-12-02; First posted 2020-01-21 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Shared Decision-making; Kidney Stone; Emergencies; Radiation Exposure; Communication
MeSH Terms: conditions — Kidney Calculi; Emergencies; Communication | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision-Making (via Decision Aid) (Experimental): The intervention is a decision aid, which both encourages and facilitates a shared decision-making conversation between the clinician and the patient. The decision aid educates patients regarding evidence-based approaches to the management of suspected kidney stones in the ED. Clinicians will receive training specific to this decision aid, though the decision aid is designed to be used with no additional training.
  Interventions: Behavioral: Decision Aid; Other: Standardized Educational Material (informational pamphlet)
- standardized educational intervention (pamphlet +usual care) (Active Comparator): The control arm will receive Usual Care and a standardized educational intervention (pamphlet). This intervention (pamphlet) contains information about kidney stones. Usual care for this clinical scenario generally involves the clinician choosing the management plan. Clinicians of subjects assigned to the usual care group will be asked to practice usual, evidence-based medical care, without shared decision-making.
  Interventions: Other: Standardized Educational Material (informational pamphlet)

INTERVENTIONS:
Behavioral: Decision Aid — Decision aid to facilitated shared decision-making
  Arms: Shared Decision-Making (via Decision Aid)
Other: Standardized Educational Material (informational pamphlet) — Pamphlet with information about kidney stones

SUMMARY:
Although a CT scan is required for some Emergency Department patients with signs and symptoms of a kidney stone, recent evidence has shown that routine scanning is unnecessary and may expose young patients to significant cumulative radiation, increasing their risk of future cancers. Shared Decision-Making may facilitate diagnostic imaging decisions that are more inline with patients' values and preferences. By comparing a shared approach to diagnostic decision-making to a traditional, physician-directed approach, this study lays the foundation for a future randomized trial that will reduce radiation exposure, improve engagement, and improve the quality and patient-centeredness of Emergency Department care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55,
2. with acute flank pain - for whom clinician believes acute flank pain may be from renal colic
3. who are deemed by the treating clinician to be at low risk for dangerous alternative diagnoses.
4. Clinician is considering imaging patient for kidney stones (any imaging)

Exclusion Criteria:

1. Recent trauma related to pain (including minor such as lifting/turning)
2. Pregnancy (previous or discovered during ED visit)
3. Recent surgical procedure on abdomen or pelvis (30d)
4. Recent urologic procedure (30d)
5. Recent childbirth (30d)
6. Signs of Systemic Infection: Fever >100.9 (101 and up), SBP <90, HR>120
7. Moderate or severe abdominal tenderness or rebound/guarding, consistently present (present for more than one exam, or present after patient treated with pain medication)
8. Second doctor's visit (ED, PCP, urgent care) for THIS episode of pain (previous similar visits ok if pain gone for >30d in between episodes) (if seen at PCP or urgent care in same day or 24 hour period, this is not an exclusion, but if seen at PCP/urgent care or ED 1-30 days prior to index visit, with same pain, excluded)
9. Known history of one kidney or other urological/renal abnormality (including neurogenic bladder, ESRD and paraplegia; or if solitary kidney discovered on US)
10. Known malignancy (any) within past year (or received treatment in the past 12 months)
11. Immunocompromised (chronic steroids, HIV, crohns, immunomodulators or severely ill chronically)
12. On anticoagulation
13. Crisis patient (behavioral health)/belligerent
14. Lacks capacity for medical decision-making
15. Unlikely to respond to follow-up calls (IVDA, homeless, no phone)
16. Clinician is concerned for alternative diagnosis requiring CT scan (appendicitis) (>5% likelihood by clinician gestalt)
17. Patient is not improving clinically and clinician is considering admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of study | Up to 12 months
  Is this study feasible? Investigators will record number of patients enrolled. An enrollment of at least three patients per month will indicate feasibility.
Fidelity | Up to 12 months
  Does the DA do what we think it is doing? Fidelity will be examined after 50 patients are enrolled: conversations between patients and clinicians will be scored for whether shared decision-making occurred. If SDM is NOT occurring in the intervention group (>75% of interactions) or IS occurring in the usual care group (>50% of interactions), fidelity will not be considered met.
Patient Knowledge | Measured at the end of the index visit. (Day 0)
  We hypothesize that the intervention group will have increased knowledge regarding radiation exposure and diagnostic options. This will be tested with a 10 question Knowledge Test developed by stakeholders for this study and delivered at the end of the index visit. The scores for this test range from 0-10 with 10 indicating higher knowledge (more correct answers)
CT scan rate | Day 0 and Day 60 (Day 60 evaluation will include all days from 0-60)
  We hypothesize that SDM will lead to a change in CT scans performed at the index visits and in the first 60 days
Radiation exposure | Day 0 and Day 60 (Day 60 evaluation will include all days from 0-60)
  We hypothesize that SDM will lead to a change in exposure to radiation. We will record radiation exposure for each CT done between day 0 and day 60, as indicated by DLP on CT reports.

SECONDARY OUTCOMES:
Patient Satisfaction | Day 0, end of visit
  Measure of satisfaction (HCAHPS measure: Provider rating where 0 = worst provider possible and 10 = best provider possible)
Patient engagement | Day 0, end of visit
  Measure of engagement: CollaboRATE 3-question measure (where 10/10 for all three is the highest score possible, and 0/0 is the lowest possible, with highest indicating better patient engagement)
Patient engagement | Day 0, end of visit
  Measure of engagement: modified CPS (Scale from 1-5, where 1 indicates the doctor made the decision, 5 indicates the patient made the decision, and 2,3, and 4 indicate levels of shared decision-making)
Patient engagement | Day 0, end of visit
  Measure of engagement: direct SDM question (Measures patients' perception of "Did SDM occur" on a likert scale of 1-7 with 1 = no and 7 = yes, and higher scores = more SDM)
Occurrence of SDM | Day 0, end of visit
  "As involved" question: "Were you as involved in today's decisions as you would have liked to be?" With three response options: Yes, No, and "There were no decisions for me to be involved in" Greater proportion of patients choosing "yes" indicates more SDM.
Occurrence of SDM | Day 0, end of visit
  Whether SDM took place from a third party observer's perspectives: OPTION-5 Score (where scale goes from 0-5, and is re-scaled to 0-100, where higher score indicates more SDM)
Overall Radiation Burden | within 60 days from index ED visit
  Radiation burden from diagnostic imaging (numeric DLP from CT reports)
Trust in physician | Day 0, end of visit
  Trust in physician scale (0-25 with 25 indicating higher trust in the physician)
ED revisits | 60 days
  Repeat visits to any Emergency Department
Safety: missed diagnosis | 60 days from index ED visit
  High Risk Diagnoses with Complications, as previously described by Smith-Bindman.
ED Length of Stay | Day 0, end of visit
  Total minutes of ED stay
Implementation Outcomes | Day 0, end of visit
  Clinician's perceptions of the conversation/intervention. We will ask about whether the clinician found the decision aid helpful, whether they would recommend it to another clinician, and whether they would use it again (likert scale 1-7 for each, with higher number indicating more acceptance/helpfulness)
Qualitative evaluation | Day 0, end of visit
  We will ask open ended questions to providers about their interaction, to ask about what went well, what did not, how else could SDM be facilitated, how this intervention would work outside of a study, what other feedback they have. This will be collected via recorded interview and open ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Schoenfeld, MD, MS, Principal Investigator — University of Massachusetts Medical School - Baystate
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan for data sharing. This could change.

REFERENCES:
- [Background] Schoenfeld EM, Poronsky KE, Westafer LM, DiFronzo BM, Visintainer P, Scales CD, Hess EP, Lindenauer PK. Feasibility and efficacy of a decision aid for emergency department patients with suspected ureterolithiasis: protocol for an adaptive randomized controlled trial. Trials. 2021 Mar 10;22(1):201. doi: 10.1186/s13063-021-05140-9. PMID 33691760